CLINICAL TRIAL: NCT05129137
Title: Pharmacokinetic Study of a Fixed Dose Combination Nefopam Hydrochloride (30 mg) / Paracetamol (500 mg) and Individual Nefopam Hydrochloride and Paracetamol Taken Alone or Concomitantly After Oral Single Dose
Brief Title: Pharmacokinetic Study of a Fixed Dose Combination Nefopam Hydrochloride (30 mg) / Paracetamol (500 mg)
Acronym: ARL/20/277
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Unither Pharmaceuticals, France (Industry)
Collaborators: Accutest Research Laboratories (I) Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: UP-CLI-2019-001
Record Dates: First submitted 2021-10-29; First posted 2021-11-22 (Actual); Results first posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Nefopam; Acetaminophen

STUDY DESIGN:
Intervention Model Description: An open-label, randomized, four-period, four treatments, cross-over trial in healthy volunteers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- FDC nefopam hydrochloride 30mg / paracetamol 500mg (Experimental): Single dose: 2 tablets
  Interventions: Drug: Combination Product: nefopam hydrochloride 30mg / paracetamol 500mg X2
- nefopam hydrochloride 30mg (Active Comparator): Single dose: 2 tablets
  Interventions: Drug: nefopam hydrochloride 30mg X2
- paracetamol 500mg (Active Comparator): Single dose: 2 tablets
  Interventions: Drug: paracetamol 500 mg X2
- nefopam hydrochloride 30mg and paracetamol 500mg (Active Comparator): Single dose: 2 tablets
  Interventions: Drug: nefopam hydrochloride 30mg X2; Drug: paracetamol 500 mg X2

INTERVENTIONS:
Drug: nefopam hydrochloride 30mg X2 — nefopam hydrochloride 30mg X2
  Arms: nefopam hydrochloride 30mg; nefopam hydrochloride 30mg and paracetamol 500mg
Drug: paracetamol 500 mg X2 — paracetamol 500 mg X2
  Other Names: acetaminophen
  Arms: nefopam hydrochloride 30mg and paracetamol 500mg; paracetamol 500mg
Drug: Combination Product: nefopam hydrochloride 30mg / paracetamol 500mg X2 — Combination Product: nefopam hydrochloride 30mg / paracetamol 500mg X2
  Arms: FDC nefopam hydrochloride 30mg / paracetamol 500mg

SUMMARY:
This study aims to assess the pharmacokinetic profile of a Fixed Dose Combination nefopam hydrochloride (30 mg) / paracetamol (500 mg) and individual components taken alone or concomitantly after oral single dose.

ELIGIBILITY:
Inclusion Criteria:

* Male and non-pregnant female human subjects, age 18 - 45 years.
* Body Mass Index between 18.5-30 Kg / m2 .
* Subjects with normal findings .
* Willingness to follow the protocol requirements

Exclusion Criteria:

* Known history of hypersensitivity to Nefopam, Paracetamol or related drugs.
* Requiring medication for any ailment having enzyme-modifying activity in the previous 28 days, prior to dosing day.
* Subjects with a history of convulsive disorders.
* Subject with a moderate or severe renal impairment
* History of cardiovascular, renal, hepatic, ophthalmic, pulmonary, neurological, metabolic, haematological, gastrointestinal, endocrine, immunological or psychiatric diseases.
* Female subjects not confirming to using birth control measures,

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2021-11-29 (Actual); Primary Completion 2021-12-27 (Actual); Study Completion 2021-12-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pramila Yadav, MS, Principal Investigator — Accutest Research Laboratories
Locations (1):
- Accutest Research Laboratories, Navi Mumbai, India

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- FDC Nefopam HCl (NEF) 30mg / APAP 500mg Then NEF 30mg + APAP 500mg Then NEF 30mg Then APAP 500mg: Participant first received 2 tablets of Investigational Medicinal Product (IMP) 08P1737F0 (Fixed Drug combination) nefopam Hydrochloride (NEF) 30mg / paracetamol (APAP) 500mg) in a fasting state. After a wash-out of 1 week, they received 2 tablets of nefopam Hydrochloride 30mg (Acupan(r)) and 2 tablets of paracetamol (Panadol(r)) 500 mg in a fasting state. After a wash-out of 1 week, they received 2 tablets of nefopam Hydrochloride 30mg (Acupan(r)) in a fasting state. After a wash-out of 1 week, they received 2 tablets of paracetamol (Panadol(r)) 500mg in a fasting state.
- NEF 30mg + APAP 500mg Then NEF 30mg Then APAP 500mg Then FDC Nefopam HCl (NEF) 30mg / APAP 500mg: Participant first received 2 tablets of nefopam Hydrochloride 30mg (Acupan(r)) and 2 tablets of paracetamol (Panadol(r)) 500mg in a fasting state. After a wash-out of 1 week, they received 2 tablets of nefopam Hydrochloride 30mg (Acupan(r)) in a fasting state. After a wash-out of 1 week, they received 2 tablets of paracetamol (Panadol(r)) 500mg in a fasting state. After a wash-out of 1 week, they received 2 tablets of IMP 08P1737F0 (FDC nefopam Hydrochloride 30mg / paracetamol 500mg) in a fasting state.
- NEF 30mg Then APAP 500mg Then FDC Nefopam HCl (NEF) 30mg Then NEF 30mg + APAP 500mg: Participant first received 2 tablets of nefopam Hydrochloride 30mg (Acupan(r)) in a fasting state. After a wash-out of 1 week, they received 2 tablets of paracetamol (Panadol(r)) 500mg in a fasting state. After a wash-out of 1 week, they received 2 tablets of IMP 08P1737F0 (FDC nefopam Hydrochloride 30mg / paracetamol 500mg) in a fasting state. After a wash-out of 1 week, they received 2 tablets of nefopam Hydrochloride 30mg (Acupan(r)) and 2 tablets of paracetamol (Panadol(r)) 500mg in a fasting state.
- APAP 500mg Then FDC Nefopam HCl (NEF) 30mg / APAP 500mg Then NEF 30mg + APAP 500mg Then NEF 30mg: Participant first received 2 tablets of paracetamol (Panadol(r)) 500mg in a fasting state. After a wash-out of 1 week, they received 2 tablets of IMP 08P1737F0 (FDC nefopam Hydrochloride 30mg / paracetamol 500mg) in a fasting state. After a wash-out of 1 week, they received 2 tablets of nefopam Hydrochloride 30mg (Acupan(r)) and 2 tablets of paracetamol (Panadol(r)) 500mg in a fasting state. After a wash-out of 1 week, they received 2 tablets nefopam Hydrochloride 30mg (Acupan(r)) in a fasting state.
Period: First Period
Arm/Group | FDC Nefopam HCl (NEF) 30mg / APAP 500mg Then NEF 30mg + APAP 500mg Then NEF 30mg Then APAP 500mg | NEF 30mg + APAP 500mg Then NEF 30mg Then APAP 500mg Then FDC Nefopam HCl (NEF) 30mg / APAP 500mg | NEF 30mg Then APAP 500mg Then FDC Nefopam HCl (NEF) 30mg Then NEF 30mg + APAP 500mg | APAP 500mg Then FDC Nefopam HCl (NEF) 30mg / APAP 500mg Then NEF 30mg + APAP 500mg Then NEF 30mg
Started | 8 | 8 | 8 | 8
Completed | 8 | 8 | 7 | 8
Not Completed | 0 | 0 | 1 | 0
Period: Second Period
Arm/Group | FDC Nefopam HCl (NEF) 30mg / APAP 500mg Then NEF 30mg + APAP 500mg Then NEF 30mg Then APAP 500mg | NEF 30mg + APAP 500mg Then NEF 30mg Then APAP 500mg Then FDC Nefopam HCl (NEF) 30mg / APAP 500mg | NEF 30mg Then APAP 500mg Then FDC Nefopam HCl (NEF) 30mg Then NEF 30mg + APAP 500mg | APAP 500mg Then FDC Nefopam HCl (NEF) 30mg / APAP 500mg Then NEF 30mg + APAP 500mg Then NEF 30mg
Started | 8 | 8 | 7 | 8
Completed | 7 | 8 | 7 | 7
Not Completed | 1 | 0 | 0 | 1
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1
Period: Third Period
Arm/Group | FDC Nefopam HCl (NEF) 30mg / APAP 500mg Then NEF 30mg + APAP 500mg Then NEF 30mg Then APAP 500mg | NEF 30mg + APAP 500mg Then NEF 30mg Then APAP 500mg Then FDC Nefopam HCl (NEF) 30mg / APAP 500mg | NEF 30mg Then APAP 500mg Then FDC Nefopam HCl (NEF) 30mg Then NEF 30mg + APAP 500mg | APAP 500mg Then FDC Nefopam HCl (NEF) 30mg / APAP 500mg Then NEF 30mg + APAP 500mg Then NEF 30mg
Started | 7 | 8 | 7 | 7
Completed | 7 | 8 | 7 | 6
Not Completed | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 1
Period: Forth Period
Arm/Group | FDC Nefopam HCl (NEF) 30mg / APAP 500mg Then NEF 30mg + APAP 500mg Then NEF 30mg Then APAP 500mg | NEF 30mg + APAP 500mg Then NEF 30mg Then APAP 500mg Then FDC Nefopam HCl (NEF) 30mg / APAP 500mg | NEF 30mg Then APAP 500mg Then FDC Nefopam HCl (NEF) 30mg Then NEF 30mg + APAP 500mg | APAP 500mg Then FDC Nefopam HCl (NEF) 30mg / APAP 500mg Then NEF 30mg + APAP 500mg Then NEF 30mg
Started | 7 | 8 | 7 | 6
Completed | 7 | 7 | 6 | 6
Not Completed | 0 | 1 | 1 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All study participants has receivent every interventions
Arm/Group | All Study Participants
Number analyzed (Participants) | 32
Age, Continuous [Least Squares Mean (Standard Deviation); unit: years] | 32.97 (6.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  India | 32

OUTCOME MEASURES:

1. Primary Outcome: Nefopam and Paracetamol Pharmacokinetic Profiles in Each Arms After Single Dose
Description: Peak Plasma Concentration (Cmax) of nefopam hydrochloride and paracetamol after single dose at different timepoints : Within 60 min before drug administration),0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 36 and 48 hours
Time Frame: up to 48 hours post dose
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | FDC Nefopam Hydrochloride 30mg / Paracetamol 500mg | Nefopam Hydrochloride 30mg | Paracetamol 500mg | Nefopam Hydrochloride 30mg and Paracetamol 500mg
Number analyzed (Participants) | 26 | 26 | 26 | 26
ng/mL
  Cmax Nefopam | 101.808 (38.283) | 114.957 (40.071) | NA (NA) — Not applicable as nefopam is not taken in this arm | 118.528 (47.616)
  Cmax Paracetamol | 13136.299 (4292.658) | NA (NA) — Not applicable as paracetamol is not taken in this arm | 21051.399 (8155.946) | 17596.380 (6431.919)

2. Primary Outcome: Nefopam and Paracetamol Pharmacokinetic Profiles in Each Arms After Single Dose
Description: Area under the plasma concentration versus time curve (AUC) of nefopam hydrochloride and paracetamol after single dose at different timepoints : Within 60 min before drug administration),0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 36 and 48 hours
Time Frame: up to 48 hours post dose
Measure: Mean (Standard Deviation); unit: ng*hr/mM
Arm/Group | FDC Nefopam Hydrochloride 30mg / Paracetamol 500mg | Nefopam Hydrochloride 30mg | Paracetamol 500mg | Nefopam Hydrochloride 30mg and Paracetamol 500mg
Number analyzed (Participants) | 26 | 26 | 26 | 26
ng*hr/mM
  AUC Nefopam | 1206.310 (541.682) | 1275.371 (511.415) | NA (NA) — Not applicable as nefopam is not taken in this arm | 1268.071 (527.581)
  AUC Paracetamol | 71402.500 (21114.375) | NA (NA) — Not applicable as paracetamol is not taken in this arm | 81877.185 (24007.993) | 78454.622 (23857.199)

3. Secondary Outcome: Paracetamol Metabolites Pharmacokinetic Profiles in Each Arms After Single Dose
Description: Peak Plasma Concentration (Cmax) of main paracetamol metabolites (Sulfate and Glucuronide) after single dose at different timepoints : Within 60 min before drug administration),0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 36 and 48 hours
Time Frame: up to 48 hours post dose
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | FDC Nefopam Hydrochloride 30mg / Paracetamol 500mg | Paracetamol 500mg | Nefopam Hydrochloride 30mg and Paracetamol 500mg
Number analyzed (Participants) | 26 | 26 | 26
ng/mL
  Cmax Paracetamol Sulfate | 6696.526 (1498.384) | 7110.342 (1664.241) | 7064.836 (1746.416)
  Cmax Paracetamol Glucuronide | 104919.677 (34090.920) | 111556.414 (38095.339) | 108171.336 (37716.515)

4. Secondary Outcome: Paracetamol Metabolites Pharmacokinetic Profiles in Each Arms After Single Dose
Description: Area under the plasma concentration versus time curve (AUC) of main paracetamol metabolites (Sulfate and Glucuronide) after single dose at different timepoints : Within 60 min before drug administration),0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 36 and 48 hours
Time Frame: up to 48 hours post dose
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | FDC Nefopam Hydrochloride 30mg / Paracetamol 500mg | Paracetamol 500mg | Nefopam Hydrochloride 30mg and Paracetamol 500mg
Number analyzed (Participants) | 26 | 26 | 26
ng*hr/mL
  AUC Paracetamol Sulfate | 53400.117 (15051.893) | 56726.962 (16795.844) | 54559.464 (16443.774)
  AUC Paracetamol Glucuronide | 848700.451 (200394.870) | 895791.865 (237880.738) | 857425.472 (209544.721)

5. Secondary Outcome: N-desmethyl-nefopam Pharmacokinetic Profiles in Each Arms After Single Dose
Description: Peak Plasma Concentration (Cmax) of N-desmethyl-nefopam after single dose at different timepoints : Within 60 min before drug administration),0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 36 and 48 hours
Time Frame: up to 48 hours post dose
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | FDC Nefopam Hydrochloride 30mg / Paracetamol 500mg | Nefopam Hydrochloride 30mg | Nefopam Hydrochloride 30mg and Paracetamol 500mg
Number analyzed (Participants) | 26 | 26 | 26
ng/mL | 31.740 (13.996) | 31.402 (13.710) | 32.279 (14.097)

6. Secondary Outcome: N-desmethyl-nefopam Pharmacokinetic Profiles in Each Arms After Single Dose
Description: Area under the plasma concentration versus time curve (AUC) of N-desmethyl-nefopam after single dose at different timepoints : Within 60 min before drug administration),0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 16, 24, 36 and 48 hours
Time Frame: up to 48 hours post dose
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | FDC Nefopam Hydrochloride 30mg / Paracetamol 500mg | Nefopam Hydrochloride 30mg | Nefopam Hydrochloride 30mg and Paracetamol 500mg
Number analyzed (Participants) | 26 | 26 | 26
ng*hr/mL | 671.457 (228.793) | 679.468 (239.053) | 692.628 (239.316)

7. Secondary Outcome: Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]
Description: Occurrence and severity of adverse events (serious and non-serious adverse events)
Time Frame: Up to 48 hours
Measure: Number; unit: event
Arm/Group | FDC Nefopam Hydrochloride 30mg / Paracetamol 500mg | Nefopam Hydrochloride 30mg | Paracetamol 500mg | Nefopam Hydrochloride 30mg and Paracetamol 500mg
Number analyzed (Participants) | 32 | 32 | 32 | 32
event | 1 | 1 | 0 | 2

ADVERSE EVENTS:
Time Frame: During the full duration of study (1 month)
Arm/Group | FDC Nefopam Hydrochloride 30mg / Paracetamol 500mg | Nefopam Hydrochloride 30mg | Paracetamol 500mg | Nefopam Hydrochloride 30mg and Paracetamol 500mg
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32 | 0/32 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32 | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 1/32 | 1/32 | 0/32 | 1/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FDC Nefopam Hydrochloride 30mg / Paracetamol 500mg (N=32) | Nefopam Hydrochloride 30mg (N=32) | Paracetamol 500mg (N=32) | Nefopam Hydrochloride 30mg and Paracetamol 500mg (N=32)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Giddiness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The CRO (ACCUTEST) shall not make any publication or communication, written or oral, in connection with the Study and the results of the Study, whether partial or final, without the prior written consent of the sponsor (UNITHER PHARMACEUTICALS) during, and following termination or expiration of this Clinical study Service Agreement

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-28): https://cdn.clinicaltrials.gov/large-docs/37/NCT05129137/Prot_SAP_000.pdf